CLINICAL TRIAL: NCT05023395
Title: Safety and Efficacy of an Investigational Medicinal Product "MEE-HU Medicus",in Combination With Antimicrobial, in Urinary Tract Infection A Randomized, Double Blind, Placebo Controlled, Multicenter Study (SEM)
Brief Title: Safety and Efficacy of MEE-HU Medicus
Acronym: (SEM)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Ahmed Ismail (Other)
Collaborators: Theodor Bilharz Research Institute (Other); The Cairo Kidney Center (Unknown); Helwan University (Other); Zagazig University (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Ahmed Ismail, Medical Research Director, Heliopolis University
Organization: Heliopolis University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00012020
Record Dates: First submitted 2021-08-23; First posted 2021-08-26 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Medicinal Product (Experimental): Patients will be assigned to receive oral MEE-HU Medicus with the empirical antibiotic. A study pharmacist will prepare visually matched packages in identical, sequentially numbered treatment packs according to a previously done computer-generated randomization list, using block randomization with variable blocks of length 4 and 6. To be dispended, in sequential order, as participants will be recruited. All participants, enrolling physicians and investigators will be blinded to the treatment allocations. Attending physicians will be responsible for enrolling the participants and ensuring that the study medications are given from the appropriate treatment pack. Selection bias is minimized by randomization, while performance bias is minimized by blinding.
  Interventions: Drug: MEE-HU Medicus
- Placebo (Placebo Comparator): Patients will be assigned to receive oral matching placebo with the empirical antibiotic. A study pharmacist will prepare visually matched packages in identical, sequentially numbered treatment packs according to a previously done computer-generated randomization list, using block randomization with variable blocks of length 4 and 6. To be dispended, in sequential order, as participants will be recruited. All participants, enrolling physicians and investigators will be blinded to the treatment allocations. Attending physicians will be responsible for enrolling the participants and ensuring that the study medications are given from the appropriate treatment pack. Selection bias is minimized by randomization, while performance bias is minimized by blinding.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MEE-HU Medicus — This investigational medicinal product (MEE-HU Medicus) is a patented mixture of amino acids and pentose sugar. The mixture according to the invention in particular is suitable as medicine for resistance-breaking of antibiotic resistances of pathogens, in particular for resistance-breaking of multiple antibiotic resistances, a method for decreasing bacterial resistance to antibiotics.
  Arms: Investigational Medicinal Product
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Primary objective: is evaluation of the investigational product's safety and evaluation of its effect, in combination with antimicrobial treatment, on urine culture (microbiological cure, no microbial growth on 24-48 hrs culture). The secondary objective: is evaluation of the investigational product's effect, in combination with antimicrobial treatment, on disease related symptoms (Clinical cure, disappearance of symptoms and signs).

DETAILED DESCRIPTION:
Design: Randomized, Double blind, Placebo controlled multicenter study. Recurrent urinary tract infection patients will blindly receive MEE-HU Medicus, or matching placebo, orally, daily, for 10 days, adjunct to the empirical antibiotic.

Population: Male and female patients over 18 years old diagnosed with recurrent urinary tract infection. Sample Size: 200 patients, 100 from each center.

ELIGIBILITY:
Inclusion Criteria:

Male and female patients over 18 years old - Symptomatic urinary tract infection (pain, dysuria, frequency, urgency, fever) confirmed by urine analysis (Pyuria, which is defined as urine WBC >10). - Negative pregnancy test and absence of vaginal discharge. - Recurrent urinary tract infection 2 times or more in the last 6 months or 3time or more in the last year. - Signed informed consent.

Exclusion Criteria Patients unable or unwilling to provide their free consent to participate in the study - Patients known or suspected to be hypersensitive to medications that will be used in the study. - Simultaneous participation in other studies. - Patients on palliative care, terminal illness. - Evidence of acute or chronic prostatitis or pyelonephritis. - History of antimicrobial use in the last 72 hrs. - Patients with renal transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-23 (Actual); Primary Completion 2024-03-24 (Estimated); Study Completion 2024-05-11 (Estimated)

PRIMARY OUTCOMES:
Complete response status | 5-7 days after completion of treatment
  Clinical cure (disappearance of symptoms and signs) and microbiological cure (negative urine culture), 5-7 days after completion of treatment.

SECONDARY OUTCOMES:
Incomplete response status | 5-7 days after completion of treatment
  Clinical cure (disappearance of symptoms and signs) with positive bacterial culture, 5-7 days after completion of treatment.

OTHER OUTCOMES:
- Failure status | 5-7 days after completion of treatment
  No clinical response, 5- days after starting of treatment.
Recurrence | 60 ±10 days from the first day of the study drug administration
  Development of new symptoms of urinary tract infection in patients with previously clinical and microbiological cure plus positive urine cultures; 60 ±10 days from the first day of the study drug administration.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo Kidney Center, Cairo
  - Theodor Bilharz Research Institute, Giza

IPD SHARING:
Plan to Share IPD: No